CLINICAL TRIAL: NCT06667973
Title: A Phase 2, Open-label, Multicentre Study Investigating Tolerability and Efficacy of Gilteritinib in Combination With Fludarabine, Cytarabine and Idarubicin (FLAI) as Induction Therapy of Newly Diagnosed Non-M3 FLT3-positive Acute Myeloid Leukemia
Brief Title: Efficacy of Gilteritinib in Combination With FLAI as Induction Therapy of FLT3-positive Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML2924
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia; FLT3 Gene Mutation; Adult AML; Diagnosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Disease | interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newly-diagnosed FLT3-positive Acute Myeloid Leukemia treated with gilteritinib (Experimental): Treatment consists in up to 2 induction cycles and up to 3 consolidation cycles:
  Induction: Patients will receive Gilteritinib 120 mg QD p.o from day 6 to 26 (21 days), in combination with FLAI induction (fludarabine 30 mg/sqm from day 1 to 5, cytarabine 2000 mg/sqm from day 1 to 5, Idarubicine 10 mg/sqm on days 1, 3, 53).
  Response will be assessed on day 28 with a bone marrow aspirate.
  * In patients not achieving CR, the second induction cycle will be identical to Induction I.
  * In patients achieving CR, a second induction cycle with ARA-C + IDA will be allowed (cytarabine 2000 mg/sqm from day 1 to 5, Idarubicine 10 mg/sqm on days 1, 3, 5), with the same schedule for Gilteritinib (day 6 to 26)
  Up to 3 consolidation cycles consisting in high dose cytarabine (1500-3000 mg/sqm bid on days 1,3,5) or intermediate in combination with Gilteritinib 120 mg QD p.o from day 6 to 26 will be allowed.
  Patients considered eligible may proceed to allo-HSCT at any time after day 28.
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — Gilteritinib fumarate is an oral, selective FLT3 and AXL inhibitor. It is a type 1 inhibitor, active against both the FLT3-ITD and FLT3-TKD mutations. Gilteritinib inhibits FLT3 receptor signaling and proliferation in cells exogenously expressing FLT3 including FLT3-ITD, FLT3-D835Y, and FLT3-ITD-D835Y, and it induces apoptosis in leukemic cells expressing FLT3-ITD.
  Gilteritinib is approved for the treatment of relpased/refractory FLT3-mutated AML after the successfull ADMIRAL trial. In the present study Gilteritinib (120 mg/die) in combination with FLAI will be tested as induction therapy in newly-diagnosed patients.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of gilteritinib as induction therapy in FLT3-positive adult acute myeloid leukemia patients. The main question it aims to answer is:

Is gilteritinib in combination to chemotherapy able to improve the complete remission rate of FLT3-positive AML?

Participants will receive up to 2 induction cycles with gilteritinib in combination with FLAI (fludarabine, cytarabine, idarubicine) and up to 3 consolidation cycles with gilteritinib and high-dose cytarabine.

DETAILED DESCRIPTION:
This is a multi-center, non-controlled, open-label, Phase 2 interventional study.

Young (≤65 years old) patients with newly diagnosed non M3, FLT3-positive acute myeloid leukemia will receive a combination of Gilteritinib and FLAI (fludarabine, high dose cytarabine and idarubicin) as induction treatment.

Gilteritinib will be administered at the standard dose of 120 mg which has already been tested in phase I combination trials. (34) Patients failing to achieve CR after first cycle may receive a second identical induction with FLAI.

Patients achieving CR after the first cycle of FLAI may receive, upon medical decision, a second induction as well, however omitting fludarabine administration (high dose cytarabine + idarubicin).

Consolidation treatment will consist in up to 3 cycles of high dose cytarabine in combination with Gilteritinib.

Transplant will be allowed in the trial for eligible patients. The primary endpoint is CR rate after first FLAI (or after second FLAI if administered).

Key secondary endpoint is MRD negativity rate after first FLAI (or after second FLAI if administered).

As the achievement of CR in AML is required for long term survival, the primary endpoint is of high clinical significance. Furthermore, given the well-known prognostic impact of MRD in CR patients, the key secondary endpoint is also highly relevant.

Planned study duration is 60 months. Patient enrollment is expected to be completed in 3 years, and the last patient enrolled will be followed-up for 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥ 18 and ≤65 years old.
2. The patient has an Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0 to 2.
3. The patient has adequate baseline organ function, including cardiac, renal, and hepatic function:

   1. Left ventricular ejection fraction (LVEF) ≥institutional lower limit of normal as measured by multigated acquisition (MUGA) scan or 2-dimensional (2-D) echocardiography (ECHO) within 21 days before start of therapy and no clinically significant abnormalities on a 12-lead electrocardiogram (ECG).
   2. ECG: QTcF≤450 male ≤480 female
   3. Serum creatinine ≤ 1.5 x ULN or an estimated glomerular filtration rate of > 50 mL/min as calculated by the Modification of Diet in Renal Disease equation.
   4. Bilirubin ≤3 times the upper limit of normal ULN mg/dL except for Gilbert's condition
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times the upper limit of normal (ULN)., except if due to leukemic involvement.
4. Patient is positive at diagnosis for FLT3 activating mutation in bone marrow or whole blood.
5. Diagnosis of untreated AML according to WHO 2016, non-APL
6. If the patient is a woman of childbearing potential (WOCBP), she must have a negative serum or urine pregnancy test at screening within 1 week before treatment.
7. The patient (male and female) agrees to use two acceptable contraceptive methods for the duration of time on the study and continue to use acceptable contraceptive methods for 6 months after the end of treatment
8. The patient has signed informed consent before initiation of any study-specific procedures or treatment.
9. The patient is able to adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment

Exclusion Criteria:

1. Patient was diagnosed as acute promyelocytic leukemia.
2. Patient has BCR-ABL-positive leukemia or chronic myelogenous leukemia in blast crisis.
3. Patient has clinically active central nervous system leukemia.
4. Patient has been diagnosed with another malignancy, unless disease-free for at least 3 years. Subjects with treated nonmelanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, papillary thyroid carcinoma, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed. Subjects with organ-confined prostate cancer with no evidence of recurrent or progressive disease are eligible if hormonal therapy has been initiated or the malignancy has been surgically removed or treated with definitive radiotherapy.
5. Patient has had major surgery within 4 weeks prior to the first study dose.
6. Patient has radiation therapy within 4 weeks prior to the first study dose.
7. Patient has congestive heart failure New York Heart Association (NYHA) class 3 or 4 or patient with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 1 month prior to study entry results in a left ventricular ejection fraction that is ≥ 45%.
8. Patient has an active uncontrolled infection.
9. Patient has active human immunodeficiency virus infection.
10. Patient has active hepatitis B or C or other active hepatic disorder. Chronic conditions previously cured or in active prophylaxis are allowed in the study
11. Patient has infections, comorbidities or any disease, condition or alteration that per judgment of the investigator may be jeopardized by therapy
12. Patients receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy with the exception of Hydroxyurea (HU) or 6-Mercaptopurine (6MP) in patients who need to continue this agent to maintain WBC count ≤10,000/mm3. HU and 6MP must be discontinued at the time of initiation of study medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate after induction | 2 months
  Number of patients who achieve a CR after course 1 or course 2 if adiministered on the total of evaluable patients

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Guolo, Principal Investigator — IRCCS Policlinico San Martino, UO Clinica Ematologica - Genova

IPD SHARING:
Plan to Share IPD: No